CLINICAL TRIAL: NCT06046937
Title: A Randomized, Double-Blind Controlled Trial of Monolaurin Ointment Versus Mupirocin Ointment of Bacterial Skin Infections Among Pediatric Patients 5-18 Years Old in Community-Based Setting
Brief Title: Monolaurin Ointment Versus Mupirocin Ointment
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Victoriano Luna Medical Center (Other Government)
Responsible Party: Principal Investigator, Wenzyl Jean Etor, Junior Consultant, Victoriano Luna Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 033/06-20
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — monolaurin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monolaurin Ointment (Experimental): treatment arm
  Interventions: Drug: Monolaurin
- Mupirocin Ointment (Active Comparator): control drug
  Interventions: Drug: Mupirocin ointment

INTERVENTIONS:
Drug: Monolaurin — applied thinly twice a day
  Other Names: Treatment Group
  Arms: Monolaurin Ointment
Drug: Mupirocin ointment — applied thinly twice a day
  Other Names: Control
  Arms: Mupirocin Ointment

SUMMARY:
Skin infection remains one of the leading causes of pediatric consults especially in developing countries like the Philippines. This common condition has not been considered a significant problem that could cause alarm as public health importance. Furthermore, due to the consideration that skin diseases are benign, not life-threatening, and low priority.

DETAILED DESCRIPTION:
The advanced technology of modern science aims to formulate a new class of antibiotics due to the emergence of antibiotic resistance in microorganisms becoming a concerning threat in the medical community. Nowadays, the use of traditional medicines derived from natural plants is in increasing demand which is geared toward going back to nature as a source of medications. 17 Recently natural plants have gained popularity in society for their medical purposes, which have important therapeutic properties that can be used in the treatment of emerging and re-emerging diseases. 17,18 Pharmaceutical companies continue to do vigorous research to discover a new antimicrobial compound with a new mechanism of action for new infectious diseases and consistently tried to find solutions to the problem of multiple resistance to the existing synthetic and conventional antimicrobial agents. Therefore, more researchers and investigators direct their attention to antimicrobial of plant origin which is found to be less in adverse reactions. 5,19 Monolaurin is a type of monoacylglycerol from lauric acid. This can be produced from varieties of oil including coconut oil. Monolaurin is included on the FDA's Generally Recognized as Safe (GRAS) list and is widely used in food manufacturing. Coconut oil naturally contains around 40-50% lauric acid, the principal compound used to make monolaurin. Studies showed, both in vitro and in vivo that monolaurin and lauric acid are very active against pathogenic bacteria. They act through several mechanisms, namely (Dayrit, 2014) (1) destruction of lipid-coated bacterial and viral cell membranes by physicochemical processes, (2) disturbances of the signal transduction and transcription in cells, (3) stabilization of the host-cells membrane (human cells). 29 Furthermore, limited clinical trials were reported on the use of monolaurin against skin infection specifically in the pediatric population. The null hypothesis of this study is that the monolaurin ointment is equivalent to mupirocin ointment in efficacy. The objective of this study was to determine the clinical efficacy of monolaurin ointment versus mupirocin ointment in the treatment of skin infections, in a community-based setting.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 5 years old to 18 years old (school-aged children)
* Subjects has infected wound (laceration, sutured wound or abrasion), impetigo and other bacterial skin infections (positive gram stain or culture)
* Subject has total skin infection rating scale score of at least 4 including pus/exudate score of at least 1
* Subject parent/legal guardian is willing and able to comply with protocol (see attached consent)
* Subject parent/legal guardian has given written informed consent or assent as applicable.
* Patient has good hygiene

Exclusion Criteria:

* Previous hypersensitivity to Mupirocin
* Secondary- infected animal/human bite or punctured wound
* Subject has a large draining abscess
* Chronic ulcerative lesion
* Other underlying skin disease
* Patient is severely malnourished
* Systemic signs and symptoms of infection
* Infection not to be appropriately treated with topical antibiotic
* Infections requires surgical intervention prior to study
* Subject received systemic antibacterial or steroid, or topical therapeutic agent within 24 hours of entry into study
* Serious underlying medical conditions/ diseases (diabetes mellitus)
* Other investigational drug within 30 days of study entry.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
success or failure of therapy | 7 days
  clinical success is determined by sufficient resolution of signs and symptoms of infection using Skin Infection Rating Scale (SIRS) Scoring: 0=absent, 1=mild, 2=moderate, 3=severe

SECONDARY OUTCOMES:
secondary outcome measure 1 | 7 days
  decrease in wound size in mm
secondary outcome measure 2 | 7 days
  post-treatment gram stain and culture result

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Sanchez, MD, Study Chair — V. Luna Medical Center
Locations (1):
- V. Luna Medical Center, Quezon City, NCR, Philippines